CLINICAL TRIAL: NCT02363218
Title: An Open-Label, Multi-Center, Single-Arm Study on Effectiveness and Safety of Stereotactic Body Radiotherapy (SBRT) Treating Hepatocellular Carcinoma Patients With CyberKnife
Brief Title: Study on Effectiveness and Safety of Hepatocellular Carcinoma Patients Treated With CyberKnife
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ping Wang
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2015-02

CONDITIONS: Liver Neoplasms
Keywords: Liver Neoplasms; Stereotactic Body Radiotherapy; CyberKnife
MeSH Terms: conditions — Liver Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CyberKnife (Experimental): Hepatocellular Carcinoma Patients Treated With CyberKnife
  Interventions: Radiation: CyberKnife

INTERVENTIONS:
Radiation: CyberKnife — Patients will undergo a CT scan with and without contrast and MRI scan for radiation treatment planning and target delineation.SBRT will be delivered on the CyberKnife with Synchrony Respiratory Tracking capabilities. The tumor will be tracked with 3 implanted fiducial seeds for targeting. Treatment will be delivered in 3 fractions within a 7 day window at the discretion of the investigator.

SUMMARY:
Study Phase: multi-institutional Phase II study Primary Objective(s): To determine overall survival for HCC patients treated with CyberKnife SBRT at 2 years.

Secondary Objective(s): 1) To determine overall survival for HCC patients treated with CyberKnife SBRT at 1 year 2) To determine local control using RECIST and EASL criteria at 1 and 2 years 3) To assess progression-free survival at 1 and 2 years 4) To assess acute and late toxicities following CyberKnife SBRT.

Hypothesis: Overall survival rate of HCC patients at one year after SBRT treatment is not less than 65%.

Study Design: Single arm study. Patients will undergo a CT scan with and without contrast and MRI scan for radiation treatment planning and target delineation.SBRT will be delivered on the CyberKnife with Synchrony Respiratory Tracking capabilities. The tumor will be tracked with 3 implanted fiducial seeds for targeting. Treatment will be delivered in 3 fractions within a 7 day window at the discretion of the investigator.

Sample size: The sample size required is 93 with a power of 90%, p=0.05, 50% response rate is considered not effective (p0) and 65% overall survival rate at 1 year (p1) is considered effectiveness of the treatment. The estimated drop-out rate is 20%, so the total sample size would be 117.

Statistical Considerations: The set of Intention-To-Treat (ITT) will be analyzed. All patients will be censored at their last visit, including the patients lost to follow-up. All patients will be followed and counted in the therapy to which they were assigned, even if they decline that therapy. Only those patients who refuse (in writing) to have their outcomes count in the study's conclusions will not be included in the analyses from that time forward; however, the follow-up data for such patients will be included up until the time they withdraw consent. Such patients will be replaced.

Baseline characteristics of patients will be presented with summary statistics. Time-to-event survival rates for OS and DFS will be estimated using the Kaplan-Meier method and presented at one and/or two years. The incidence of acute and late toxicities will be presented in tabular form on both a per-patient and per-event basis.

DETAILED DESCRIPTION:
Indication: Hepatocellular carcinoma (HCC) is the third most deadly cancer in the world. It is primarily seen in areas where hepatitis is endemic, such as Asia, but other risk factors include alcoholic cirrhosis.

Surgical resection and/or transplantation remain the only curative options. However, more than 80% of patients present with unresectable disease. For these patients with unresectable tumors, a variety of treatment options are available, including transarterial chemoembolization (TACE), radiofrequency ablation (RFA), radioactive microspheres, microwave coagulation, laser-induced thermotherapy, and percutaneous alcohol injection, all of which have similar survival rates. Stereotactic body radiotherapy (SBRT) for unresectable HCC is a relatively new treatment option made available because of significant improvements in diagnostic imaging and radiation delivery techniques. Although follow-up is limited, results show encouraging local control rates.

The investigators propose to conduct a Phase II study assessing the efficacy and safety of CyberKnife SBRT for the treatment of HCC.

Summary of Subject Eligibility Criteria:

Inclusion Criteria

1. Confirmed hepatocellular carcinoma according to one of three EASL criteria:

   * Histopathology
   * Two radiographic techniques (out of US, MRI, CT, Angiography) that confirm a lesion >2 cm with arterial hypervascularization
   * One radiographic technique that confirms a lesion >2 cm with arterial hypervascularization and an AFP>400 ng/mL
2. Unifocal liver tumors not to exceed 5 cm in greatest axial dimension. Multifocal lesions will be restricted to a maximum of 3 lesions with a maximum lesion size of 3 cm for each lesion, that can be treated within a single target volume within the same liver segment as long as the dose constraints to normal tissue can be met.
3. Volumn of uninvolved liver >750 cc
4. Hepatic lesion in patients for whom surgical resection is not possible or patients who refuse surgery.
5. Eastern Clinical Oncology Group (ECOG) performance status 0, 1 or 2 (Appendix I)
6. Patients with liver disease classified as Child Pugh class A
7. Life expectancy >6 months
8. Age > 18 years old
9. Albumin > 2.5 g/dL
10. Total Bilirubin < 3 mg/dL
11. INR <1.5
12. Transaminases (SGOT and SGPT) no more than 3 times the upper limit of normal
13. Creatinine < 2.0 mg/dL
14. Both men and women and members of all races and ethnic groups are eligible for this study
15. Ability of the research subject or authorized legal representative to understand and the willingness to sign a written informed consent document Exclusion Criteria

1. Prior surgery, chemotherapy or radiation for the liver tumor 2. Prior radiotherapy to the upper abdomen 3. Prior RFA or liver transplant 4. Tumors greater than 5 cm in greatest axial dimension 5. Child B status 6. Contraindication to receiving radiotherapy 7. Active gastrointestinal bleed within 2 weeks of study enrollment 8. Clinically significant ascites refractory to medical therapy 9. Women who are pregnant 10. Administration of any systemic chemotherapy within the last 6 months 11. Presence of multifocal lesions located in different lobes of the liver or extrahepatic metastases 12. Portal vein thrombus 13. Participation in another concurrent treatment protocol Intervention and Mode of Delivery: CyberKnife SBRT - External photon radiation. Procedure is outpatient. Synchrony Respiratory Tracking System Duration of Intervention and Evaluation: The duration of treatment will be 1 week.. The follow-up period will be for 3 years following completion of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed hepatocellular carcinoma according to one of three EASL criteria:

   * Histopathology
   * Two radiographic techniques (out of US, MRI, CT, Angiography) that confirm a lesion >2 cm with arterial hypervascularization
   * One radiographic technique that confirms a lesion >2 cm with arterial hypervascularization and an AFP>400 ng/mL
2. Unifocal liver tumors not to exceed 5 cm in greatest axial dimension. Multifocal lesions will be restricted to a maximum of 3 lesions with a maximum lesion size of 3 cm for each lesion, that can be treated within a single target volume within the same liver segment as long as the dose constraints to normal tissue can be met.
3. Volumn of uninvolved liver >750 cc
4. Hepatic lesion in patients for whom surgical resection is not possible or patients who refuse surgery.
5. Eastern Clinical Oncology Group (ECOG) performance status 0, 1 or 2 (Appendix I)
6. Patients with liver disease classified as Child Pugh class A
7. Life expectancy >6 months
8. Age > 18 years old
9. Albumin > 2.5 g/dL
10. Total Bilirubin < 3 mg/dL
11. INR <1.5
12. Transaminases (SGOT and SGPT) no more than 3 times the upper limit of normal
13. Creatinine < 2.0 mg/dL
14. Both men and women and members of all races and ethnic groups are eligible for this study
15. Ability of the research subject or authorized legal representative to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Prior surgery, chemotherapy or radiation for the liver tumor
2. Prior radiotherapy to the upper abdomen
3. Prior RFA or liver transplant
4. Tumors greater than 5 cm in greatest axial dimension
5. Child B status
6. Contraindication to receiving radiotherapy
7. Active gastrointestinal bleed within 2 weeks of study enrollment
8. Clinically significant ascites refractory to medical therapy
9. Women who are pregnant
10. Administration of any systemic chemotherapy within the last 6 months
11. Presence of multifocal lesions located in different lobes of the liver or extrahepatic metastases
12. Portal vein thrombus
13. Participation in another concurrent treatment protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | Two years

SECONDARY OUTCOMES:
Overall survival rate | One year
Local Control rate | Two years
Progression-free survival | One-Two Years

CONTACTS AND LOCATIONS:
Overall Officials: PING WANG, MD.PHD, Principal Investigator — Tianjin Medical University Institute & Hospital
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Background] Bruix J, Sherman M; Practice Guidelines Committee, American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma. Hepatology. 2005 Nov;42(5):1208-36. doi: 10.1002/hep.20933. No abstract available. PMID 16250051
- [Background] Bruix J, Hessheimer AJ, Forner A, Boix L, Vilana R, Llovet JM. New aspects of diagnosis and therapy of hepatocellular carcinoma. Oncogene. 2006 Jun 26;25(27):3848-56. doi: 10.1038/sj.onc.1209548. PMID 16799626
- [Background] Blomgren H, Lax I, Naslund I, Svanstrom R. Stereotactic high dose fraction radiation therapy of extracranial tumors using an accelerator. Clinical experience of the first thirty-one patients. Acta Oncol. 1995;34(6):861-70. doi: 10.3109/02841869509127197. PMID 7576756
- [Background] Cardenes HR, Price TR, Perkins SM, Maluccio M, Kwo P, Breen TE, Henderson MA, Schefter TE, Tudor K, Deluca J, Johnstone PA. Phase I feasibility trial of stereotactic body radiation therapy for primary hepatocellular carcinoma. Clin Transl Oncol. 2010 Mar;12(3):218-25. doi: 10.1007/s12094-010-0492-x. PMID 20231127
- [Background] Fuss M, Salter BJ, Herman TS, Thomas CR Jr. External beam radiation therapy for hepatocellular carcinoma: potential of intensity-modulated and image-guided radiation therapy. Gastroenterology. 2004 Nov;127(5 Suppl 1):S206-17. doi: 10.1053/j.gastro.2004.09.035. PMID 15508086
- [Background] Herfarth KK, Hof H, Bahner ML, Lohr F, Hoss A, van Kaick G, Wannenmacher M, Debus J. Assessment of focal liver reaction by multiphasic CT after stereotactic single-dose radiotherapy of liver tumors. Int J Radiat Oncol Biol Phys. 2003 Oct 1;57(2):444-51. doi: 10.1016/s0360-3016(03)00586-8. PMID 12957256
- [Background] Herfarth KK, Debus J, Lohr F, Bahner ML, Rhein B, Fritz P, Hoss A, Schlegel W, Wannenmacher MF. Stereotactic single-dose radiation therapy of liver tumors: results of a phase I/II trial. J Clin Oncol. 2001 Jan 1;19(1):164-70. doi: 10.1200/JCO.2001.19.1.164. PMID 11134209
- [Background] Katz AW, Carey-Sampson M, Muhs AG, Milano MT, Schell MC, Okunieff P. Hypofractionated stereotactic body radiation therapy (SBRT) for limited hepatic metastases. Int J Radiat Oncol Biol Phys. 2007 Mar 1;67(3):793-8. doi: 10.1016/j.ijrobp.2006.10.025. Epub 2006 Dec 29. PMID 17197128
- [Background] Kavanagh BD, Scheftera TE, Wersall PJ. Liver, renal, and retroperitoneal tumors: stereotactic radiotherapy. Front Radiat Ther Oncol. 2007;40:415-426. doi: 10.1159/000106051. PMID 17641524
- [Background] Lax I, Blomgren H, Naslund I, Svanstrom R. Stereotactic radiotherapy of malignancies in the abdomen. Methodological aspects. Acta Oncol. 1994;33(6):677-83. doi: 10.3109/02841869409121782. PMID 7946448
- [Background] Mendez Romero A, Wunderink W, Hussain SM, De Pooter JA, Heijmen BJ, Nowak PC, Nuyttens JJ, Brandwijk RP, Verhoef C, Ijzermans JN, Levendag PC. Stereotactic body radiation therapy for primary and metastatic liver tumors: A single institution phase i-ii study. Acta Oncol. 2006;45(7):831-7. doi: 10.1080/02841860600897934. PMID 16982547
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Estimating the world cancer burden: Globocan 2000. Int J Cancer. 2001 Oct 15;94(2):153-6. doi: 10.1002/ijc.1440. No abstract available. PMID 11668491
- [Background] Schefter TE, Kavanagh BD, Timmerman RD, Cardenes HR, Baron A, Gaspar LE. A phase I trial of stereotactic body radiation therapy (SBRT) for liver metastases. Int J Radiat Oncol Biol Phys. 2005 Aug 1;62(5):1371-8. doi: 10.1016/j.ijrobp.2005.01.002. PMID 16029795
- [Background] Takeda A, Takahashi M, Kunieda E, Takeda T, Sanuki N, Koike Y, Atsukawa K, Ohashi T, Saito H, Shigematsu N, Kubo A. Hypofractionated stereotactic radiotherapy with and without transarterial chemoembolization for small hepatocellular carcinoma not eligible for other ablation therapies: Preliminary results for efficacy and toxicity. Hepatol Res. 2008 Jan;38(1):60-9. doi: 10.1111/j.1872-034X.2007.00084.x. Epub 2007 May 15. PMID 17506837
- [Background] Tse RV, Hawkins M, Lockwood G, Kim JJ, Cummings B, Knox J, Sherman M, Dawson LA. Phase I study of individualized stereotactic body radiotherapy for hepatocellular carcinoma and intrahepatic cholangiocarcinoma. J Clin Oncol. 2008 Feb 1;26(4):657-64. doi: 10.1200/JCO.2007.14.3529. Epub 2008 Jan 2. PMID 18172187
- [Background] Wada H, Takai Y, Nemoto K, Yamada S. Univariate analysis of factors correlated with tumor control probability of three-dimensional conformal hypofractionated high-dose radiotherapy for small pulmonary or hepatic tumors. Int J Radiat Oncol Biol Phys. 2004 Mar 15;58(4):1114-20. doi: 10.1016/j.ijrobp.2003.08.012. PMID 15001252